CLINICAL TRIAL: NCT00500253
Title: Assessment of Utility of Exhaled Nitric Oxide Measurement for Treatment Monitoring in Children With Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RNN-56-07-KE
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: exhaled nitric oxide; asthma; children; inhaled glucocorticosteroids
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): children with asthma with FeNO monitored treatment (study group)
  Interventions: Device: exhaled nitric oxide measurement; Procedure: bronchial hyperresponsiveness with methacholine (PC20M)
- 2 (Other): group of children with treatment monitored by GINA's grade of disease clinical control (control group)
  Interventions: Procedure: bronchial hyperresponsiveness with methacholine (PC20M); Procedure: symptom score diary (according to 2007 GINA guidelines)

INTERVENTIONS:
Device: exhaled nitric oxide measurement — exhaled nitric oxide measurement
  Other Names: exhaled nitric oxide measurement (Sievers FeNO analyzer)
  Arms: 1
Procedure: bronchial hyperresponsiveness with methacholine (PC20M) — bronchial hyperresponsiveness with methacholine (PC20M)
  Other Names: PC20M Jaeger APS system
Procedure: symptom score diary (according to 2007 GINA guidelines) — symptom score diary (according to 2007 GINA guidelines)
  Arms: 2

SUMMARY:
The aim of this study is to assess the utility of exhaled nitric oxide measurement (FeNO) in treatment monitoring in children with asthma.

According to the aim of the study following assumptions are formulated:

1. Comparison of annual cumulative steroid dose, number of bronchodilator doses taken, number of asthma exacerbation, number of hospitalisation due to asthma, between group of children with asthma with FeNO monitored treatment (study group), and group of children with treatment monitored by GINA's grade of disease clinical control (control group)
2. Assessment of corelation of FeNO (ppb) with symptom score (points)and lung function (FEV1)
3. Comparison of values of non-specific bronchial hyperresponsiveness with methacholine (PC20M)between both study groups after 12. months of treatment.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic disease worldwide, imposing a substantial social burden on both children and adults.

What needs to be kept in mind, especially in assessing treatment effect of allergic inflammation in children with asthma, is that symptom score and spirometry measures have limitations, mainly their subjectivity (symptom scores), wide variability, and lack of stability in short time period (symptom scores and spirometry measures).

Monitoring allergic inflammation in the course of asthma in children with exhaled nitric oxide measurement (FeNO) may allow to titrate the dose of inhaled glucocorticosteroids more precisely, depending on individual patients requirements.

The aim of this study is to assess the utility of FeNO in treatment monitoring in children with asthma.

According to the aim of the study following assumptions are formulated:

1. Comparison of annual cumulative steroid dose, number of bronchodilator doses taken, number of asthma exacerbation, number of hospitalisation due to asthma, between group of children with asthma with FeNO monitored treatment (study group), and group of children with treatment monitored by GINA's grade of disease clinical control (control group)
2. Assessment of corelation of FeNO (ppb) with symptom score (points)and lung function (FEV1)
3. Comparison of values of non-specific bronchial hyperresponsiveness with methacholine (PC20M)between both study groups after 12. months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* FeNO values above the norm for age and inadequate asthma control (based GINA guidelines)

Exclusion Criteria:

* presence of other perennial and seasonal allergies
* presence of other chronic diseases
* excluded medications: systemic glucocorticosteroids 3 months before enrollment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Control of the disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sołoniewicz, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Lodz, Poland, Lodz, Poland